CLINICAL TRIAL: NCT02955134
Title: Follow-up Study of Chinese Medicine for the Treatment of Chronic Atrophic Gastritis Based on Histological Evaluation
Brief Title: The Study of Chinese Medicine for the Treatment of Chronic Atrophic Gastritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing University of Chinese Medicine (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Shaanxi Hospital of Traditional Chinese Medicine (Other); Gansu Provincial Hospital (Other); Tianjin Nankai Hospital (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Hebei Hospital of Traditional Chinese Medicine (Unknown); Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital (Unknown); Shanxi Province hospital Research Institute of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); Shanghai University of Traditional Chinese Medicine (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201507001-09
Record Dates: First submitted 2016-10-28; First posted 2016-11-04 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Chronic Atrophic Gastritis
Keywords: central blinded histological assessment; traditional Chinese medicine intervention; biological specimen banks
MeSH Terms: conditions — Gastritis, Atrophic | interventions — hydrotalcite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese medicine prescription (Experimental): On the basis of symptomatic treatment of Talcid® and Compound Azimtamide Entieric-coated Tablets,patients in experimental group use the traditional Chinese medicine application prescription.
  Interventions: Drug: Talcid®; Drug: Chinese medicine prescription; Drug: Compound Azimtamide Entieric-coated Tablets
- placebo (Placebo Comparator): On the basis of symptomatic treatment of Talcid® and Compound Azimtamide Entieric-coated Tablets,patients in placebo group use the simulate granule of traditional Chinese medicine application prescription.
  Interventions: Drug: Talcid®; Drug: Placebo; Drug: Compound Azimtamide Entieric-coated Tablets

INTERVENTIONS:
Drug: Talcid® — Talcid® is allowed to be taken when patients feel stomach pain, acid reflux or heartburn. Continuous taking time should not exceed one week.
Drug: Chinese medicine prescription — The Chinese medicine application prescription is composed of pinellia 9g, radix scutellariae 10g, rhizoma coptidis 8g, rhizoma zingiberis 10g, radix curcumae 10g, rhizoma atractylodis 10g, roasted bighead atractylodes rhizome 10g, radix astragali 15g, spreading hedyotis herb 20g, scutellariae barbatae 20g, salvia miltiorrhiza bge 10g, the stem of noble dendrobium 10g, radix pseudostellariae 10g, fructus aurantii immaturus 10g, cortex magnoliae officinalis 10g, rhizoma curcumae 10g, ginger 3g, jujube 6g.
  Patients take 200ml each time, twice a day. Treatment duration are 24 weeks.
  Arms: Chinese medicine prescription
Drug: Placebo — The placebo is simulate granule of Chinese medicine application prescription. Patients take 200ml each time, twice a day. Treatment duration are 24 weeks.
  Arms: placebo
Drug: Compound Azimtamide Entieric-coated Tablets — Compound Azimtamide Entieric-coated Tablets are qualified by China Food and Drug Administration. These tablets are allowed to be taken when patients feel fullness, belching or anorexia. Continuous taking time should not exceed one week.

SUMMARY:
The purpose of this study is to evaluate efficacy of Chinese medicine treatment for chronic atrophic gastritis. It is a multi-center, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
A prospective, double-blind, randomized, placebo-controlled, multi-center trial is carried out in this study.The sample size is 468 patients ( 312 in treatment group, 156 in control group). The investigators will screen the patients for inclusion according to the inclusion and exclusion criteria. All patients detect of H.pylori, undergo upper digestive endoscopy and biopsies for histological investigation. Patients infected of H.pylori must receive H.pylori eradication therapy under the guidance of Kyoto global consensus report on H.pylori gastritis. Then they are assigned to treatment group or control group with an allocation ratio of 2:1. Patients intreatment group take the traditional Chinese medicine prescription, while the control group take simulate granule of the prescription. Both two groups are under symptomatic treatment. Treatment duration lasts 24 weeks. Investigators also follow up another 24 weeks. Histological changes are used as the primary outcome index. Endoscopy findings, symptoms are assessed. Serum level of pepsinogen and patient-reported outcome instrument are also administered during the study. All biopsy specimens are collected to build the biological specimen bank. Central blinded histological assessment (Histological diagnosis is determined independently by three experienced pathologists who are blinded to the information of the patients.) are used to insure the accuracy and consistency. Tele-medicine and information management system is established to help achieve follow-up interviews.

Random numbers are generated by SAS 9.4 software. The subjects, caregivers, investigators and outcomes assessors in this study are all blinded.

ELIGIBILITY:
Inclusion criteria

1. Patients diagnosed with chronic atrophic gastritis.
2. Patients whose pathological diagnosis was atrophy (reduction glands) of mild/moderate grade，with or without intestinal metaplasia, with or without mild/moderate dysplasia.
3. Aged between 40 to 65 years old, male or female.
4. Patients who agree to participate in the clinical study through informed consent.
5. Local residents ensuring regular treatment and follow-up.
6. Not taking aspirin, warfarin and other anticoagulants and those without coagulation disorders.

Exclusion criteria

1. Autoimmune gastritis.
2. The combined gastric and duodenal ulcers, upper gastrointestinal bleeding.
3. Dysplasia of severe degree,or suspicious of gastric malignancy.
4. Serious comorbidities of heart, lung, liver, kidney or blood system (such as cardiac function above grade II, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than 1.5 times the upper limit of normal, creatinine (Cr) greater than the upper limit of normal and so on) or having a life-threatening illness .
5. Psychiatric disorders or a history of alcohol or drug abuse.
6. Pregnant or lactating women.
7. Allergic to the trial drug.
8. Patients judged inappropriate to participate in the trial by investigators.
9. Patients enrolled in another clinical trial last two months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change of histological score | Change from baseline histological score at 6 months and 1 year
  Gastric mucosa samples are subsequently evaluated according to updated Sydney system with the degree of H.pylori density, polymorphonuclear neutrophil activity, chronic inflammation, glandular atrophy, and intestinal metaplasia classified as: 0,'absent'; 2, 'mild'; 4, 'moderate'; and 6, 'marked'. Grade of histological gastritis is evaluated with this score 0, 2, 4, and 6. Dysplasia was assessed according to the revised Vienna classification, scored as 0 (absent), 2 (mild), 4 (moderate), or 6 (marked).
Change of symptoms score | Change from baseline symptoms score at 6 months and 1 year
  Symptoms of dyspepsia, regurgitation and defecation are assessed for severity and frequency at enrollment in every interview during the study.For each symptom, the scores are calculated by multiplying frequency by severity.
  All symptom scores are added to define the total symptom score.

SECONDARY OUTCOMES:
Change of endoscopic atrophy | Change from baseline endoscopic atrophy at 6 months and 1 year
  Endoscopic atrophy are defined using an endoscopicatrophic border scale previously reported by Kimura and Takemoto. This scale correlates with histological results and includes the following classifications: 1 close-type, when the atrophic border remains on the lesser curvature of the stomach; 2 open-type, when the atrophic border extends along the anterior and posterior walls of the stomach and is not associated with the lesser curvature of the stomach. Close-type and open-type atrophy are further classified as none (C0), mild (C1, 2),moderate (C3, O1), and severe (O2, 3) atrophy. In this study, atrophy grade are also scored as C0: 0, C1: 1, C2: 2, C3:3, O1: 4, O2: 5, and O3: 6 respectively, with 0 representing an absence of atrophy and 6 indicating severe atrophy.
Change of OLGA stages. | Change from baseline at 6 months and 1 year
  Three expert GI pathologists, who are blinded for the endoscopic findings, independently assessed all biopsy specimens of the surveillance endoscopy. The type and grade of the different stages of changes are classified according to the updated Sydney system and scored as 0 (absent), 1 (mild), 2(moderate), or 3 (marked) by using the Sydney system visual analog scale. On the basis of the standardized sites, the gastritis stages areassess according to the OLGA.
Change of OLGIM stages. | Change from baseline endoscopic atrophy at 6 months and 1 year
  Three expert GI pathologists, who are blinded for the endoscopic findings, independently assessed all biopsy specimens of the surveillance endoscopy. The type and grade of the different stages of changes are classified according to the updated Sydney system and scored as 0 (absent), 1 (mild), 2(moderate), or 3 (marked) by using the Sydney system visual analog scale. On the basis of the standardized sites, the gastritis stages areassess according to the OLGA.

OTHER OUTCOMES:
Change of serum level of pepsinogen | Change from baseline serum level of pepsinogen at 6 months and 1 year
  serum level of pepsinogen Ⅰ in ng/ml， pepsinogen Ⅱ in ng/ml, pepsinogen Ⅰ/pepsinogen Ⅱ
Patient-Reported Outcome Instrument developed by our research group. | through study completion, an average of 1 month
  The Patient-Reported Outcome Scale is developed by our research group，and this scale involves the dimensions of patients' reaction in physical, psychological and social function.
Blood routine tests | up to 24 weeks
  Blood routine tests including
Electrocardiogram | up to 24 weeks
Renal function | up to 24 weeks
  BUN, Cr
Liver function | up to 24 weeks
  ALT, AST
Stool routine tests | up to 24 weeks
Urine routine tests | up to 24 weeks
Adverse events | up to 24 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wei, Ph.D, Principal Investigator — Wangjing Hospital of China Academy of Chinese Medical Sciences
Locations (13):
- China (13):
  - Beijing Hospital of Traditional Chinese Medicine Affiliated to Capital Medical University, Beijing
  - Wangjing Hospital of China Academy of Chinese Medical Sciences, Beijing
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing
  - Guangdong Provincial TCM Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou
  - GanSu Provincial Hospital of Traditional Chinese Medicine, Lanzhou
  - Yueyang Hospital of Integrated Traditional Chinese Medicine and Western Medicine, Affiliated Hospital of Shanghai University of Traditional Chinese Medicine, Shanghai
  - Liaoning Hospital of TCM, Shenyang
  - Hebei Hospital of TCM, Shijiazhuang
  - Shanxi province hospital of traditional Chinese medicine, Taiyuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin
  - Tianjin Nankai Hospital, Tianjin
  - Shanxi Traditional Chinese Medicine Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided